CLINICAL TRIAL: NCT02421055
Title: Longitudinal Phenotyping of Bariatric Surgery Patients
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 15SM2479
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: Bariatric Surgery; Gastric Bypass; Sleeve Gastrectomy; Gastroplasty
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Serum, urine and stool preoperatively and at 3 months and 1 year postoperatively.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Roux-en-Y Gastric Bypass
  Interventions: Procedure: Laparoscopic Roux-en-Y Gastric Bypass
- Group 2: Sleeve Gastrectomy
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-Y Gastric Bypass
  Groups: Group 1
Procedure: Laparoscopic Sleeve Gastrectomy
  Groups: Group 2

SUMMARY:
Recent studies have shown that bacteria within the gut play an important role in diabetes improvement after bariatric (weight-loss) surgery. Bariatric surgery fundamentally changes the environment within the gut, which results in changes to the makeup of the trillions of bacteria living within it. These changes in the gut bacteria can affect the body in a number of complex ways, which we are only just beginning to understand. For example, gut bacteria breakdown food we are unable to absorb ourselves, leading to altered sugar levels and can release molecules that act to reduce appetite.

In this study we aim to find out how bariatric surgery changes the gut bacteria and how this leads to weight loss and improvement of diabetes. With this understanding we hope to discover potential targets for future treatments, such as identifying beneficial bacteria that could be supplemented with probiotics in patients.

Additionally, although highly successful, up to 30% of obese patients do not undergo improvement of their diabetes after bariatric surgery. We aim to identify molecules within the patient's blood or urine that are able to predict the likely chance a patient will undergo improvement in their diabetes after bariatric surgery to help clinicians select patients most likely to benefit.

DETAILED DESCRIPTION:
This study aims to assess how the gut microbiome affects the host phenotype following bariatric surgery through altered gut microbiome-host co-metabolism. The secondary objective is to identify novel biomarkers for the preoperative prognostication of T2DM remission following bariatric surgery.

The study will longitudinally phenotype obese diabetics and non-diabetics undergoing Roux-en-Y Gastric Bypass or Sleeve Gastrectomy surgery. Patients will be assessed preoperatively and at 3 months and 1 year postoperatively. Clinical measures recorded will include; 1) anthropometric & physiological measurements, 2) demographic details, 3) biochemical parameters including HbA1c, 4) anti-hyperglycaemic and other medication use, 5) co-morbidity status and 6) dietary choices through 24hr dietary recall questionnaires.

Blood, urine and stool samples will be collected at the above time points. Changes to the microbiome will be assessed using metagenomic sequencing. Global metabonomic profiles of serum, urine and faecal water will be generated using 1H-NMR. Further targeted analyses of bile acid and short-chain fatty acid profiles will be performed using LC-MS / GC-MS.

The study will utilise multivariate statistical analysis techniques to identify metabolic pathways altered following intervention, and novel host-microbiome co-metabolism pathways that impact upon phenotype. A supervised multivariate analysis, mapping T2DM outcomes to metagenomic and metabonomic data will be performed with the aim of identifying novel preoperative biomarkers that are able to prognosticate T2DM resolution following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI>30kg/m2)
* Type 2 Diabetes Mellitus and non-diabetic
* Failure of efforts at lifestyle modification and dieting
* Fitness for anaesthesia and procedure
* Willingness to comply with the trial protocol

Exclusion Criteria:

* Previous bariatric surgery
* Pregnancy or intention to become pregnant during trial period
* Lack of capacity to consent
* Previous major abdominal surgery (Small or large bowel resection, stomach, liver, pancreatic or splenic surgery. Does not include patients who have previously had an appendicectomy, cholecystectomy or hernia repair).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with obesity undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Darzi, MB, BCh, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Weight Centre, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants consented to give serum samples only, others were able to give complete sets of serum, 24-hour urine and stool, as detailed below.
Groups:
- Pre-operative Only: Recruited patients that did not undergo RYGB or VSG procedures
- Roux-en-Y Gastric Bypass (RYGB): Participants who underwent RYGB procedure
- Vertical Sleeve Gastrectomy (VSG): Participants who underwent VSG procedure
Period: Overall Study
Arm/Group | Pre-operative Only | Roux-en-Y Gastric Bypass (RYGB) | Vertical Sleeve Gastrectomy (VSG)
Started | 34 | 50 | 74
Pre-operative Serum Sample (Minimum) | 34 | 50 | 74
Pre-operative Complete Sample Set (Complete sample set of serum, 24-hour urine and stool) | 23 | 22 | 36
Post-operative Serum Sample (Minimum) | 0 | 23 | 26
Post-operative Complete Sample Set (Complete sample set of serum, 24-hour urine and stool) | 0 | 13 | 14
Completed (Clinical data collected at pre-operative and post-operative time points) | 0 | 50 | 74
Not Completed | 34 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with at least one pre-operative serum sample
Groups:
- Roux-en-Y Gastric Bypass (RYGB): 50 participants gave pre-operative serum samples prior to undergoing RYGB. 23 participants underwent RYGB and gave serum samples pre and 3-months post-operatively.
  13 of these gave complete sample sets of serum, 24-hour urine and stool pre and 3-months post-operation.
- Vertical Sleeve Gastrectomy (VSG): 74 participants gave pre-operative serum samples prior to undergoing VSG. 26 participants underwent VSG and gave serum samples pre and 3-months post-operatively.
  14 of these gave complete sample sets of serum, 24-hour urine and stool pre and 3-months post-operation.
- Total: Total of all reporting groups
Arm/Group | Roux-en-Y Gastric Bypass (RYGB) | Vertical Sleeve Gastrectomy (VSG) | Total
Number analyzed (Participants) | 50 | 74 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.54 (11.04) | 44.01 (11.91) | 45.03 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 49 | 90
  Male | 9 | 25 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50 | 74 | 124
Weight (Kg) [Mean (Standard Deviation); unit: Kg] | 120.86 (20.17) | 133.6 (30.35) | 128.14 (27.29)
BMI (kg/m2) [Mean (Standard Deviation); unit: Kg/m2] | 44.43 (5.69) | 47.12 (8.99) | 46.03 (7.91)
Diabetes Status [Count of Participants; unit: Participants]
  Type 2 Diabetes (T2D) | 27 | 24 | 51
  Impaired Glucose Tolerence (IGT) | 7 | 13 | 20
  Non-diabetic | 16 | 37 | 53
HBA1c [Mean (Standard Deviation); unit: mmols/mol] | 52.24 (17.66) | 45.41 (12.82) | 48.16 (15.27)
Metformin use [Count of Participants; unit: Participants] | 26 | 22 | 48
Insulin use [Count of Participants; unit: Participants] | 10 | 5 | 15
Duration of T2D (years) [Mean (Standard Deviation); unit: years] — Population: T2D participants only
  years
    number analyzed (Participants) | 27 | 24 | 51
    (all) | 7.96 (7.03) | 7.75 (8.47) | 7.86 (7.66)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Diabetes Remission at 3 Months
Description: Participants with HbA1c <6% (42mmol/mol), off anti-diabetic medication, at 3 months
Time Frame: 3 months
Population: Participants with complete follow up data
Measure: Count of Participants; unit: Participants
Groups:
- Roux-en-Y Gastric Bypass: Participants who underwent Roux-en-Y Gastric Bypass
- Vertical Sleeve Gastrectomy: Participants who underwent Vertical Sleeve Gastrectomy
Arm/Group | Roux-en-Y Gastric Bypass | Vertical Sleeve Gastrectomy
Number analyzed (Participants) | 18 | 16
Participants | 8 | 5

2. Secondary Outcome: Partial Diabetes Remission
Description: HbA1c <6.5% (48mmol/mol), off anti-diabetic medication, at 3 months. (Includes participants with complete remission).
Time Frame: 3 months
Population: Participants with complete follow up data
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: Vertical Sleeve Gastrectomy
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 18 | 16
Participants | 9 | 6

3. Secondary Outcome: HbA1c Improvement
Description: Reduction in HbA1c at 3 months
Time Frame: 3 months
Population: Participants attending follow up
Measure: Mean (Standard Deviation); unit: mmols/mol
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 44 | 67
mmols/mol | 12.0 (11.98) | 7.53 (10.18)

4. Secondary Outcome: Weight Loss
Description: Weight loss at 3 months
Time Frame: 3 months
Population: Participants attending follow up
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 44 | 67
Kg/m2 | 24.13 (9.13) | 24.00 (7.94)

5. Secondary Outcome: BMI Reduction
Description: BMI reduction at 3 months
Time Frame: 3 months
Population: Participants attending follow up
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 44 | 67
Kg/m2 | 8.87 (2.99) | 8.51 (2.62)

6. Secondary Outcome: Complete Diabetes Remission
Description: HbA1c <6% (42mmol/mol), off anti-diabetic medication, at 1 year
Time Frame: 1 year
Population: Participants with complete follow up data
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 15 | 12
Participants | 10 | 4

7. Secondary Outcome: Partial Diabetes Remission
Description: HbA1c <6.5% (48mmol/mol), off anti-diabetic medication, at 1 year. (Includes participants with complete diabetes remission).
Time Frame: 1 year
Population: Participants with complete follow up data
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 15 | 12
Participants | 10 | 5

8. Secondary Outcome: HbA1c Improvement
Description: Reduction in HbA1c at 1 year
Time Frame: 1 year
Population: Participants attending follow up
Measure: Mean (Standard Deviation); unit: mmols/mol
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 36 | 57
mmols/mol | 13.72 (13.71) | 6.88 (10.19)

9. Secondary Outcome: Weight Loss
Description: Weight loss at 1 year
Time Frame: 1 year
Population: Participants attending follow up
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 36 | 57
Kg | 37.53 (11.36) | 35.23 (12.98)

10. Secondary Outcome: BMI Reduction
Description: BMI reduction at 1 year
Time Frame: 1 year
Population: Participants attending follow up
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 36 | 57
Kg/m2 | 13.8 (3.69) | 13.02 (5.54)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious, and other adverse events were not monitored/assessed. None occurred as a result of this observational study.
Groups:
- Pre-operative Samples Only: Recruited patients that did not undergo RYGB or VSG procedures
- Roux-en-Y Gastric Bypass: Participants who underwent RYGB
- Vertical Sleeve Gastrectomy: Participants who underwent VSG
Arm/Group | Pre-operative Samples Only | Roux-en-Y Gastric Bypass | Vertical Sleeve Gastrectomy
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/50 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Complete sets of serum, 24-hour urine and faeces were not collected from all participants. Details are described in baseline group descriptions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT02421055/Prot_SAP_000.pdf